CLINICAL TRIAL: NCT00570791
Title: The Effect of Central Corneal Thickness On Intraocular Pressure Measurements With the Goldman Applanation Tonometer, Ocular Blood Flow Pneumatonometer,Tono Pen,Pascal Dynamic Contour Tonometer, and Schiotz Tonometer
Brief Title: Effect of Central Corneal Thickness On IOP Using Various Tonometers
Acronym: CCT
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0441-04-FB
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Intraocular Pressure
Keywords: Cornea; Tonometers; Goldmann applanation; Tonopen; Shiotz; Pneumatonometer
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Effect of age on intraocular pressure: Correlation between age and IOP with GAT compared to other tonometers.
  Interventions: Device: Tonometer
- Effect of CCT and IOP: Correlation between CCT and IOP among all tonometers
  Interventions: Device: Tonometer

INTERVENTIONS:
Device: Tonometer — Tonometer devices used to measure IOP: Pascal Dynamic Contour Tonometer, Goldman Applanation Tonometer, Tono Pen, Reichart pneumatonometer, Langham Ocular Blood Flow, Schiotz Tonometer and ICare tonometer

SUMMARY:
The primary purpose of this study is to evaluate the effects of ocular physical properties on intraocular pressure (IOP) measurements in eyes with healthy corneas using the following instruments to measure IOP: Goldmann applanation tonometer, pneumotonometer, ocular blood flow pneumotonometer, Tono-Pen, Pascal Dynamic Contour Tonometer and the Schiotz Tonometer. Ocular physical properties to be evaluated are:varying (CCT), corneal curvature (CC), axial length, anterior chamber depth and scleral rigidity. The secondary purpose of this is to determine if there is a correlation between CCT and other ocular properties, and which instruments that measure these other ocular properties are most affected by CCT.

DETAILED DESCRIPTION:
Accurate estimation of intraocular pressure is an essential aspect in the diagnosis and management of glaucomatous eye disease. Glaucoma is a progressive optic neuropathy and a leading cause of blindness in the United States. In glaucoma, vision is lost through apoptosis (programmed cell death) of retinal ganglion cells, a type of cell in the retina that transmits visual information to the brain. Diagnosis of glaucoma is usually based on a combination of progressive, characteristic vision loss (measured using visual field testing) and progressive optic nerve head damage (as detected through dilated fundus examinations or disc photography). While a high pressure inside the eye (ocular hypertension, OHT) is not sufficient for a diagnosis of glaucoma, it is the greatest single risk factor for disease onset.

For decades, the gold standard for intraocular pressure measurement has been the Goldmann applanation tonometer. The Goldmann tonometer is calibrated based on a central corneal thickness of 500 micrometers. But, it is known that CCT varies between individuals and even between individual eyes. The various central corneal thicknesses (CCT)s are thought to influence the accuracy of IOP measurements and thus the diagnosis, screening, and treatment of patients with glaucoma. A study performed by Copt (1999) showed that ocular hypertensive patients have relatively thick corneas and normal tension glaucoma patients have relatively thin corneas. Thus it is thought that a thicker cornea creates falsely high IOP readings and a thinner cornea creates falsely low IOP readings. This was followed by a study performed by Lleo et al (2003) which showed that applanation tonometry and CCT positively correlated in normal eyes. More recently the following studies have also found a positive correlation between CCT and tonometry: Lui et al (2005), Tonnu et all (2005), Pourjavan et al (2005), Doyle et al (2005), Gunvant et al (2005), Brunsini et al (2005) and Rask et al (2005).

To further evaluate the effect of CCT on IOP measurement, the method and instruments used to measure IOP were compared. In a clinical setting IOP's are measured by four instruments, Goldmann applanation tonometer, ocular blood flow pneumatonometer, pneumatonometer or Tono-Pen. Singh et al (2001) concluded that the effect of central corneal thickness on Goldmann applanation tonometry accuracy appears not to be clinically relevant. However, Bhan et al (2002) showed that in eyes with normal corneas, the ocular blood flow pneumatonometer appears to be more affected by variation in CCT than the Goldmann tonometer, and the Tono-Pen is least affected by CCT. A limitation of this study is that corneal curvature (a measure of astigmatism) was not performed prior to measuring IOP. High amounts of astigmatism can impact IOP readings obtained from the Goldmann tonometer.

The PASCAL Dynamic Contour Tonometer is a new digital tonometer that provides a direct trans-corneal measurement of IOP and is sensitive enough to detect the ocular pulse amplitude (OPA) due to the patient's heartbeat. Supposedly, when using the principle of contour matching instead of applanation, the PASCAL eliminates the systematic errors inherent in all previous tonometers, such as the influence of corneal thickness and rigidity. Ku et al (2005) demonstrated that the Pascal tonometer was effective in reducing corneal thickness bias during IOP measurements.

It has long been thought that there is a significant positive correlation of scleral rigidity to IOP, thus with increasing pressure in the eye, a resulting increase in rigidity is noted. (1960). A study completed by Pallikaris et al. (2005) investigated a possible correlation of rigidity to other ocular found no correlation between the two.

The effect of CCT on IOP measurement is a clinical concern as erroneous IOP measurements may lead to misdiagnosis. The purpose of this study is to evaluate whether IOP measurements by Goldmann applanation, pneumotonometryocular blood flow pneumotonometry, y, Tono-Pen and the PASCAL Dynamic Contour Tonometer are affected by central corneal thickness, and if so, to what extent.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19.
* Patients may or may not be on IOP lowering medication.

Exclusion Criteria:

* History of baseline corneal disease including but not limited to: Fuchs' Dystrophy, Keratoconus, Iridocorneal Endothelial Syndrome, Lattice Dystrophy, Map-Dot- Fingerprint Dystrophy, or a history of Stevens-Johnson Syndrome.
* Wears hard or rigid contact lenses.
* History of inflammatory eye disease.
* History of ocular trauma within the past 6 months.
* History of ocular infection within the last 3 months.
* Any abnormality preventing reliable IOP readings.
* Subject has demonstrated potential for non-compliance with the study protocol (e.g. dosing schedule, visit schedule, or study procedures).
* History of severe hypersensitivity to topical fluorescein.
* Pregnant or breast feeding women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinic Patients, City Residents
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2005-06-29 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-11-01 (Actual)

PRIMARY OUTCOMES:
Eye pressure | one - two hours
  Measured pressure in participants' eyes with six different tonometers

CONTACTS AND LOCATIONS:
Overall Officials: Carol B Toris, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Department of Ophthalmolgy and Visual Sciences, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska